CLINICAL TRIAL: NCT01205178
Title: A Phase I Study to Investigate the Hemolytic Potential of Tafenoquine in Healthy Subjects With Glucose-6-phosphate Dehydrogenase Deficiency and the Safety and Tolerability of Tafenoquine in Acute Plasmodium Vivax Malaria Patients With Glucose-6-phosphate Dehydrogenase Deficiency
Brief Title: G6PD (Glucose-6-phosphate Dehydrogenase) Study to Evaluate Hemolysis Potential of TFQ (Tafenoquine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 110027
Record Dates: First submitted 2010-03-18; First posted 2010-09-20 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Chloroquine; Primaquine; tafenoquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tafenoquine (Active Comparator): Tafenoquine, TQ is an 8-aminoquinoline (8-AQ) antimalarial drug being developed for the radical cure of acute P. vivax malaria. Chloroquine will be given for the first 3 days in second and third part of this study to treat Malaria.
  Interventions: Drug: Chloroquine; Drug: Tafenoquine
- Chloroquine (Active Comparator): Dose for first 3 days for Part B & C of the study
  Interventions: Drug: Chloroquine
- Primaquine (Active Comparator): once daily for first 14 days
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Chloroquine — The current gold standard for radical cure of P. vivax malaria in many areas of the world is chloroquine (CQ); typically 600 mg day 1, 600 mg day 2, 300 mg day 3 for clearance of the acute parasitemia. After this Tafenoquine will be given and subject will be followed up.
  Arms: Chloroquine; Tafenoquine
Drug: Primaquine — Primaquine (PQ) is another 8 aminoquinoline drug available for Malaria treatment
  Arms: Primaquine
Drug: Tafenoquine — Once daily on Day 1 only. For Part B and C of this study Chloroquine will be given to treat Malaria
  Arms: Tafenoquine

SUMMARY:
SB-252263 (Tafenoquine, TQ) is an 8-aminoquinoline (8-AQ) antimalarial drug being developed by GlaxoSmithKline (GSK), the U.S. Army Medical Research and Materiel Command (USAMRMC) and Medicines for Malaria Venture (MMV). TQ is currently being developed for the radical cure of acute P. vivax malaria in combination with standard doses of CQ, which is 1500 mg over 3 days.

The current gold standard for radical cure of P. vivax malaria in many areas of the world is chloroquine (CQ) for clearance of the acute parasitemia immediately followed by primaquine (PQ) to clear the liver stages of the parasite and prevent disease relapse. The 8-AQ class of drugs, including PQ, is hemolytic in subjects with glucose-6-phosphate dehydrogenase (G6PD) deficiency. The current study will identify a dose of TQ within the target efficacious dose range that has a hemolytic effect similar to or less than PQ 15 mg OD x 14 days (i.e. ≤ 25-30% hemoglobin decline in WHO class III G6PD-deficient subjects).

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* The subject is between 18 and 45 years of age, inclusive
* A female is eligible to enter and participate in this study if she is non-pregnant, non-lactating and if she is of:
* Non-child bearing potential defined as:
* Is post-menopausal (12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH >40mIU/mL)
* Is pre-menopausal and has had a hysterectomy or a bilateral oophorectomy (removal of the ovaries) or a bilateral tubal ligation with medical report verification.
* Child-bearing potential, has a negative urine pregnancy test at screening, and agrees to comply with one of the following during the treatment stage of the study and for a period of 90 days after stopping study drug:
* Use of oral contraceptive, either combined or progestogen alone, in combination with a barrier method (e.g., condom or diaphragm)
* Use of an intrauterine device with a documented failure rate of less than 1% per year
* Double barrier method consisting of spermicide with either condom or diaphragm.
* Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female
* Complete abstinence from intercourse for 2 weeks prior to administration of study drug, throughout the study and for a period of 90 days after stopping study drug.
* A signed and dated informed consent is obtained from the subject or the subject's legal representative prior to screening.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* WHO class III G6PD-deficiency or G6PD-normal status must be documented by enzyme activity and cytochemical staining. G6PD genotype must confirm WHO class III G6PD deficiency or G6PD-normal status prior to TQ dosing in all parts of the study (i.e., P. vivax infected subjects may commence CQ therapy whilst the cytochemical staining, enzyme activity and G6PD genotype are being determined).

Supplemental Inclusion Criteria for Part A: Healthy volunteers Inclusion criteria 1-7 above AND

* Subject is female
* For G6PD-deficient subjects (WHO class III variant), subject must be heterozygous with 40-60% normal RBCs by cytochemical staining method. For G6PD-normal subjects, subject must have >90% normal RBCs by cytochemical staining method.

Supplemental Inclusion Criteria for Part B: P. vivax patients Inclusion criteria 1-7 above AND

* Subject is female
* Positive blood smear for P. vivax with parasite density >500 and <200,000/µl
* For G6PD-deficient subjects (WHO class III variant), subject must be heterozygous with 40-60% normal RBC by cytochemical staining method. For G6PD-normal subjects, subject must have >90% normal RBCs by cytochemical staining method.

Supplemental Inclusion Criteria for Part C: P. vivax patients Inclusion criteria 1-7 above AND

* Positive blood smear for P. vivax with parasite density >500 and <200,000/µl
* For G6PD-deficient subjects (WHO class III variant), subject is a homozygous female or a hemizygous male. For G6PD-normal subjects, subject must have >90% normal RBCs by cytochemical staining method

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Clinically significant illness (intercurrent illness e.g. pneumonia, pre-existing condition e.g. renal disease, malignancy or conditions that may affect absorption of study medication e.g. severe diarrhea or any signs of malnutrition as defined clinically, and clinical signs and symptoms of vascular disease (e.g. cardiac, CNS, diabetes, hyperlipidemia, etc.).
* Any clinically relevant biological or physical abnormality found or reported at screening which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study. These abnormalities may be identified on the screening history and physical or laboratory examination, 12-lead electrocardiogram (ECG).
* Mixed malaria infections by Giemsa smear.
* Female subjects who are pregnant, lactating or unwilling/unable to comply with recognized contraceptive methods during the treatment stage of the study and for a period of 90 days after stopping study drug.
* Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
* History of hemoglobinopathy (e.g. sickle-cell disease, hereditary spherocytosis, thalassemias, hemoglobin M, etc.); or current or past history of methemoglobinemia or methemoglobin percentage above 3%.
* History of porphyria
* History of psoriasis
* History of allergy to tafenoquine, chloroquine, primaquine, mefloquine or any other 4- or 8-aminoquinolines.
* Subject has taken other anti-malarials (e.g., mefloquine, primaquine, chloroquine) within the past 60 days by history.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Donation of blood in excess of 500mL within 56 days prior to dosing study drug.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (one drink = five ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* History of illicit drug abuse within 6 months of the study.
* Heparin sensitivity (if heparin is used to maintain intravenous catheter patency).
* QTc interval >450 msec at screening Supplemental Exclusion Criteria for Part A: Healthy volunteers Exclusion criteria 1-16 above AND
* Baseline Hgb <12 g/dL (or Hct <36%). Value to be verified by conducting two measurements (single blood draw).
* Use of prescription or non-prescription drugs, vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 28 days prior to the first dose of study medication. Unless in the opinion of the investigator and sponsor the medication will not interfere with study procedures or compromise safety. By exception, the subject may take paracetamol or acetaminophen (≤2 grams/day) up to 48 hours prior to the first dose of study medication.

Supplemental Exclusion Criteria for Parts B and C: P. vivax patients

Exclusion criteria 1-16 above AND Laboratory criteria for exclusion are:

* platelets <50,000/µL
* WBC <2000/µL
* Calculated creatinine clearance (CrCl) <50ml/min by Cockcroft-Gault formula:
* Men: CrCl = (140 - age) x weight(kg)/(72 x SCr*)
* Woman: CrCl = [(140 - age) x weight(kg)/(72 x SCr*)] x 0.85

  *SCr= serum creatinine
* ALT or AST >2 times upper limit of the reference range
* Total bilirubin level >1.5 times upper limit of the reference range at screening.
* Screening Hgb <11 g/dL (or Hct <33%). Value to be verified by conducting two measurements (single blood draw).

Subjects who have taken or will likely require the use of medications from the prohibited medication list which include the following classes:

* Histamine-2 blockers and antacids
* Drugs with hemolytic potential
* Drugs known to prolong the QTc interval

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2009-07-02 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2013-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, and hemolytic potential of TQ in G6PD-deficient female healthy volunteers compared with G6PD-normal female healthy volunteers. This will be done by measuring maximum absolute decline in Haemoglobin from baseline | 2 years

SECONDARY OUTCOMES:
Maximum absolute decline in Hgb (or Hct) from baseline for TQ in G6PD-deficient healthy volunteers compared to G6PD-normal healthy volunteers. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Tak

REFERENCES:
- See also: Results for study 110027 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110027?search=study&search_terms=110027#rs